CLINICAL TRIAL: NCT05465733
Title: A Prospective, Single-arm, Single-center Clinical Trial of Envafolimab as First-line Replacement Maintenance in Advanced NSCLC
Brief Title: First-line Replacement Maintenance of Envafolimab in Advanced NSCLC
Acronym: NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.XJTU1AF2022LSK-263
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-03

CONDITIONS: Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab (Experimental)
  Interventions: Drug: Envafolimab;Pemetrexed

INTERVENTIONS:
Drug: Envafolimab;Pemetrexed — single agent, 300mg Q3W IH until disease progressed,The duration of treatment with Envafolimab should not exceed 2 years.

SUMMARY:
This study is a single-center, prospective, single-arm phase II clinical study. For newly-treated patients with advanced NSCLC with negative driver gene and positive PD-L1 expression, those patients who did not progress after 4-6 cycles of PD-1 or PD-1 combined with chemotherapy standard treatment, after signing the informed consent form, were screened to meet the criteria for inclusion and exclusion. Standard, will receive Envafolimab combined with chemotherapy/Envafolimab single-agent first-line maintenance therapy until disease progression, withdrawal of informed consent, initiation of other anti-tumor therapy, death, or other protocol-specified conditions that should be discontinued Circumstances, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up;
2. Age 18-75 years old;
3. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC);
4. Patients with non-small cell lung cancer (NSCLC) who have received PD-1 or PD-1 combined with chemotherapy and have not progressed in previous first-line therapy;
5. According to the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1), at least one lesion that can be measured by imaging. Lesions located in the field of previous radiotherapy can be regarded as measurable lesions if they are confirmed to have progressed;
6. An archived tumor tissue sample or newly obtained (no anti-tumor therapy since biopsy) core or tumor foci (no prior radiotherapy) excisional biopsy has been provided. Formalin-fixed and paraffin-embedded (FFPE) tissue blocks are preferred over sections. The newly obtained biopsy tissue is superior to the archived tissue, and the tissue sample is detected by immunohistochemistry for PD-L1 ≥ 1%;
7. ECOG score 0-1 points;
8. Expected survival time ≥ 3 months;
9. Sufficient organ function, subjects should meet the following laboratory indicators:

(1) The absolute value of neutrophils (ANC) is ≥1.5x109/L without the use of granulocyte colony-stimulating factor in the past 14 days; (2) Platelets ≥100×109/L without platelet transfusion or thrombopoietin use in the past 14 days; (3) Hemoglobin>9g/dL without blood transfusion or erythropoietin in the past 14 days; (4) Total bilirubin ≤ 1.5 × upper limit of normal (ULN); or total bilirubin > ULN but direct bilirubin ≤ ULN (5) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are ≤2.5×ULN (patients with liver metastases are allowed ALT or AST ≤5×ULN); (6) Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥60 ml/min; (7) Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; for patients receiving anticoagulation therapy, PT/INR is within the required treatment criteria; (8) Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled; (9) Myocardial enzyme spectrum is within the normal range (if the investigators comprehensively judge that the simple laboratory abnormality does not have clinical significance, it is also allowed to be included in the group); 10. For female subjects of childbearing age, a negative urine or serum pregnancy test should be performed within 3 days prior to receiving the first dose of study drug (Day 1 of Cycle 1). If a urine pregnancy test result cannot be confirmed negative, a blood pregnancy test is required. Women of non-reproductive age are defined as having been postmenopausal for at least 1 year, or have undergone surgical sterilization or hysterectomy; 11.If there is a risk of conception, all subjects (whether male or female) are required to use an annual failure rate of less than 1 throughout the treatment period up to 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapy drug) % of contraception.

Exclusion Criteria:

1. Patients with known EGFR sensitive mutations or ALK rearrangements;
2. Patients who have received first-line standard treatment and progressed in the past;
3. Subjects with active central nervous system (CNS) metastasis, if the subject's CNS metastasis can be adequately treated, and the subject's neurological symptoms can return to baseline levels at least 2 weeks before enrollment treatment-related residual signs or symptoms), can participate in the study. In addition, the subject must also be a corticosteroid-free subject or receive a stable or tapering dose of ≤10 mg/day of prednisone (or equivalent);
4. Received systemic systemic treatment of Chinese patent medicines with anti-lung cancer indications or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use for controlling pleural effusion) within 2 weeks before the first administration;
5. Currently participating in interventional clinical research treatment, or have received other investigational drugs or used investigational device treatment within 4 weeks before the first dose;
6. Active autoimmune disease requiring systemic treatment (such as the use of disease-modifying drugs, glucocorticoids or immunosuppressants) has occurred within 2 years before the first dose. Replacement therapy (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) is not considered systemic therapy;
7. Are receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose of the study; Note: Physiological doses of glucocorticoids (≤10 mg/day prednisone or equivalent) are allowed;
8. Those who are known to be allergic to the active ingredients or excipients of the study drugs such as envolimab and pemetrexed;
9. Pregnant or lactating women;
10. Has not sufficiently recovered from toxicity and/or complications from any intervention (ie, ≤ Grade 1 or reached baseline, excluding fatigue or alopecia) prior to initiating treatment;
11. Known history of human immunodeficiency virus (HIV) infection (ie HIV 1/2 antibody positive);
12. Untreated active hepatitis B (defined as HBsAg positive and the detection of HBV-DNA copy number greater than the upper limit of the normal value of the laboratory department of the research center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load <1000 copies/ml (200 IU/ml) before the first dose, subjects should receive anti-HBV therapy throughout the study treatment period to avoid viral reactivation;
2. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), prophylactic anti-HBV treatment is not required, but viral reactivation needs to be closely monitored; 13. Active HCV infected subjects (HCV antibody positive and HCV-RNA level higher than the detection limit); 14. Received live vaccine within 30 days before the first dose (cycle 1, day 1); Note: Injected inactivated virus vaccine against seasonal influenza within 30 days prior to the first dose is permitted; however, intranasal live attenuated influenza vaccine is not permitted.

15. Presence of any serious or uncontrolled systemic disease such as:

1. There are significant abnormalities in the rhythm, conduction or morphology of the resting ECG, and the symptoms are severe and difficult to control, such as complete left bundle branch block, second-degree heart block, ventricular arrhythmia or atrial fibrillation;
2. Unstable angina pectoris, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) classification ≥ grade 2;
3. Myocardial infarction occurred within 6 months before enrollment;
4. Unsatisfactory blood pressure control (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);
5. There is a history of non-infectious pneumonia requiring glucocorticoid treatment within 1 year before the first administration, or there is currently clinically active interstitial lung disease;
6. Active pulmonary tuberculosis;
7. There is an active or uncontrolled infection that requires systemic treatment;
8. Clinically active diverticulitis, abdominal abscess, and gastrointestinal obstruction;
9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
10. Poor control of diabetes (fasting blood glucose (FBG) > 10mmol/L);
11. Urine routine indicates urine protein ≥++, and 24-hour urine protein quantification >1.0 g;
12. Patients with mental disorders and unable to cooperate with treatment; 16. Medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the results of the trial, prevent the subjects from participating in the research throughout the study, or the investigator considers other circumstances that are not suitable for inclusion or have other potential risks and are not suitable to participate in this research. .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 3-year
  time from the randomization to the first disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No